CLINICAL TRIAL: NCT01311713
Title: An Open-Label Study to Determine the Maximum Tolerated Dose of the PARP Inhibitor CEP-9722 When Administered as a Single Agent in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study to Determine the Maximum Tolerated Dose of the PARP Inhibitor CEP-9722 in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C9722/2051; 2010-023657-12 (EudraCT Number)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumors
Keywords: cancer; tumors; PARP
MeSH Terms: conditions — Neoplasms | interventions — CEP-9722; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- CEP-9722 Dose 1 QD (Experimental): Participants will receive Dose 1 of CEP-9722 tablet once daily (QD) orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 1 BID (Experimental): Participants will receive Dose 1 of CEP-9722 tablets twice daily (BID) orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 2 BID (Experimental): Participants will receive Dose 2 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 3 BID (Experimental): Participants will receive Dose 3 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 4 BID (Experimental): Participants will receive Dose 4 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 5 BID (Experimental): Participants will receive Dose 5 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722
- CEP-9722 Dose 6 BID (Experimental): Participants will receive Dose 6 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
  Interventions: Drug: CEP-9722

INTERVENTIONS:
Drug: CEP-9722 — CEP-9722 will be administered per dose and schedule specified in the arm description.
  Other Names: poly ADP ribose polymerase Inhibitor

SUMMARY:
CEP-9722 is an inhibitor of poly-adenosine diphosphate (ADP) ribose polymerase -1 and -2 (PARP). The primary purpose of this study is to (Part 1) determine the maximum tolerated dose (MTD) of CEP-9722 administered daily to participants with advanced or metastatic solid tumors, (Part 2) to evaluate the safety and tolerability of that dose, and to investigate whether CEP-9722 has antitumor activity as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically confirmed, locally advanced or metastatic solid tumor considered incurable and unresponsive to standard therapies.
* The participant has disease progression following at least 1 prior standard chemotherapy regimen.
* The participant is a man or woman at least 18 years of age.
* The participant has a European Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* The participant has a life expectancy of 12 weeks or more.
* The participant has adequate hematologic function as evidenced by:
* absolute neutrophil cell (ANC) count 1.5 x10^9/liter (L) or more
* hemoglobin 10 grams (g)/deciliter (dL) or more
* platelets 100 x 10^9/L or more
* The participant has adequate hepatic function as evidenced by:
* total bilirubin 1.5 times the upper limit of normal (ULN) or less, unless secondary to Gilbert's disease (any Gilbert's disease must be documented, and bilirubin must be 3 times the ULN or less.)
* alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase of 2.5 times ULN or less
* The participant has adequate renal function as defined by creatinine of less than 1.5 times ULN or less.
* The participant must take precautions to not become pregnant or produce offspring. Women must be of non-childbearing potential (surgically sterile or postmenopausal for at least 12 months, confirmed by follicle-stimulating hormone [FSH] >40 IU/L) or agree to use a medically accepted method of contraception for the duration of the study and 90 days after treatment. Men must be surgically sterile or agree to use a medically accepted method of contraception for the duration of the study and 90 days after treatment. Acceptable methods of contraception include abstinence, barrier method with spermicide (excluding cervical cap and sponge), intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* Written informed consent is obtained.
* In Part 2: In addition to the criteria above, participants should have documented deficiencies of DNA repair pathways, such as BRCA1/2, or have prostate, breast, or gastric cancer and ability to provide fresh or archived tumor specimens.

Exclusion Criteria:

* Other than malignancy, the participant has any serious or uncontrolled surgical, medical, or psychiatric history that could pose an unacceptable health risk to the participant, prevent compliance with study procedures, or compromise the study integrity, including, but not limited to the following:

  1. recent history of cardiac ischemic disease (acute myocardial infarction within 6 months, unstable angina)
  2. cardiac arrhythmia that is uncontrolled or that requires medication
  3. recent transient ischemic attack or stroke (within 6 months) or residual dysfunction from stroke
  4. history of seizure disorder (part 1 only)
  5. clinically significant pulmonary disease (eg, fibrosis on chest x-ray or significant dyspnea as assessed by investigator)
  6. poorly controlled hypertension (systolic >140 millimeters of mercury (mm Hg) or diastolic >90 mm Hg)
  7. uncontrolled active infection within the past 7 days
  8. poorly controlled diabetes mellitus as assessed by investigator
  9. recent major surgery (within 4 weeks prior to study day 1) or minor surgery (within 2 weeks prior to study day 1)
* The participant has previously received a PARP inhibitor.
* The participant has received antitumor therapy or other investigational agent within 4 weeks (with the exception of LHRH therapy in participants with prostate cancer) or nitrosourea therapy within 6 weeks.
* The participant has clinically symptomatic brain metastases or required treatment for brain metastases within 4 weeks (stable sequelae acceptable if treatment has been completed).
* The participant has residual adverse events of greater than grade 1 severity from prior radiotherapy or chemotherapy agents.
* The participant has known immunodeficiency virus (HIV) infection, acute or chronic hepatitis B infection,or hepatitis C infection.
* The participant is a pregnant or breast-feeding woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The participant has medical or surgical gastrointestinal history that would interfere with the absorption of study drug.
* The participant requires treatment with a proton pump inhibitor or H2 antagonist or has taken a proton pump inhibitor or H2 antagonist within 4 days before CEP-9722 administration.
* The participant has risk factors for Torsades de Pointes as follows:
* history of Long QT syndrome or unexplained syncope
* history of congestive heart failure (New York Heart Association class III or IV)
* concomitant treatment with medication known to prolong QT/QTc interval
* QTc greater than 450 milliseconds (msec) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2013-10-16 (Actual); Study Completion 2013-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (4):
- United States (4):
  - Teva Investigational Site 1, Aurora, Colorado
  - Teva Investigational Site 3, Detroit, Michigan
  - Teva Investigational Site 4, St Louis, Missouri
  - Teva Investigational Site 2, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts: Part 1 (to determine the maximum tolerated dose [MTD] of single agent oral CEP-9722) and Part 2 (to evaluate the safety and tolerability of the MTD of CEP-9722 identified in Part 1). The study was stopped before reaching its primary objective of determining the MTD of CEP-9722. The lowest dose of CEP-9722 administered was 150 milligrams (mg) and the highest dose was 1000 mg.
Groups:
- CEP-9722 Dose 1 QD: Participants received Dose 1 of CEP-9722 tablet once daily (QD) orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 1 BID: Participants received Dose 1 of CEP-9722 tablets twice daily (BID) orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 2 BID: Participants received Dose 2 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 3 BID: Participants received Dose 3 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 4 BID: Participants received Dose 4 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 5 BID: Participants received Dose 5 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 6 BID: Participants received Dose 6 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
Period: Overall Study
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Started | 3 | 7 | 9 | 6 | 5 | 6 | 9
Received at Least 1 Dose of Study Drug | 3 | 7 | 8 | 6 | 5 | 6 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 9 | 6 | 5 | 6 | 9
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1 | 2
Not completed — Disease progression | 3 | 4 | 3 | 2 | 4 | 4 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Stopped taking study medication | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Enrolled but not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other than specified | 0 | 1 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of CEP-9722.
Groups:
- CEP-9722 Dose 1 QD: Participants received Dose 1 of CEP-9722 tablet QD orally with a standard meal for up to 6 cycles of 28 days each.
- CEP-9722 Dose 1 BID: Participants received Dose 1 of CEP-9722 tablets BID orally with a standard meal for up to 6 cycles of 28 days each.
- Total: Total of all reporting groups
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID | Total
Number analyzed (Participants) | 3 | 7 | 8 | 6 | 5 | 6 | 9 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (7.00) | 63.9 (6.04) | 57.0 (13.85) | 60.2 (7.83) | 50.6 (12.84) | 59.3 (16.32) | 57.2 (13.33) | 57.8 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 6 | 5 | 4 | 4 | 8 | 34
  Male | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 7 | 5 | 4 | 5 | 6 | 37
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 6 | 7 | 6 | 3 | 5 | 5 | 35
  Race: Black | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 6
  Race: Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race: Other | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Tolerated Dose (MTD) of Oral CEP-9722
Description: MTD was defined as the highest dose level with 0 or 1 participant experiencing a dose-limiting toxicity (DLT) during cycle 1. DLT was defined as any adverse event (AE) that was considered by the investigator as related or potentially related to CEP-9722 as follows: 1) hematologic: grade 4 hematologic adverse events, grade 3 or greater febrile neutropenia, grade 3 thrombocytopenia lasting 7 days or more, grade 3 thrombocytopenia with bleeding; 2) nonhematologic: grade 3 or 4 nonhematologic AEs; grade 4 vomiting or diarrhea; grade 3 nausea, vomiting, or diarrhea that persisted for 48 hours or more despite optimal medical intervention; QTcF (QTc by Fridericia's cube root formula) greater than 500 milliseconds (msec) (confirmed by a repeat measurement on the same visit). During Cycle 1 of Part 1, any toxicity possibly related to treatment with CEP-9722 that caused a cumulative interruption of dosing for 7 or more days was considered dose limiting.
Time Frame: Cycle 1 (28 days)
Population: The MTD determination set included all participants who received at least 1 dose of the study drug during the first cycle. In addition, any participant who experienced a drug related DLT during cycle 1 was considered evaluable regardless of the number of doses received.
Measure: Number; unit: milligram (mg)
Groups:
- Overall Population: Participants received CEP-9722 orally with a standard meal for up to 6 cycles of 28 days each.
Arm/Group | Overall Population
Number analyzed (Participants) | 44
milligram (mg) | NA — The MTD was not calculated. The study was terminated due to pharmacokinetic variability and lack of clinical activity.

2. Primary Outcome: Part 2: Number of Participants With Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to 8 months
Population: Part 2 of the study was not conducted, hence there were no analyses for any of the Part 2 outcome measures.
Arm/Group | Overall Population
Number analyzed (Participants) | 0

3. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of CEP-8983 (the Active Moiety of CEP-9722)
Time Frame: Predose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, and 12 hours postdose on Days 1 and 15 of Cycle 1
Population: The pharmacokinetic (PK) analysis set included participants for whom at least 1 PK parameter can be calculated. Here, 'number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Number analyzed (Participants) | 3 | 7 | 9 | 6 | 5 | 6 | 9
nanograms (ng)/milliliter (mL)
  Cycle 1 Day 1 | 285.7 (282.03) | 695.6 (425.14) | 1585.4 (921.33) | 1808.8 (921.42) | 3136.8 (2387.63) | 4306.2 (1177.27) | 4121.1 (1729.05)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 6 | 6 | 5 | 3 | 6
  Cycle 1 Day 15 | 271.7 (264.19) | 575.5 (346.35) | 888.7 (407.73) | 1492.7 (881.44) | 2332.4 (990.45) | 2753.3 (537.66) | 4679.8 (2047.07)

4. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Time of Last Measurable Drug Concentration (AUC0-t) of CEP-8983 (the Active Moiety of CEP-9722)
Time Frame: Predose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, and 12 hours postdose on Days 1 and 15 of Cycle 1
Population: The PK analysis set included participants for whom at least 1 PK parameter can be calculated. Here, 'number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Number analyzed (Participants) | 3 | 7 | 9 | 6 | 5 | 6 | 9
ng*hours/mL
  Cycle 1 Day 1 | 1309.0 (1550.61) | 3416.3 (2813.31) | 10050.0 (6100.96) | 13996.2 (8845.35) | 16527.4 (9711.19) | 40914.7 (14594.45) | 49332.9 (26717.97)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 6 | 6 | 5 | 3 | 6
  Cycle 1 Day 15 | 930.3 (1320.83) | 2758.5 (1353.95) | 3507.7 (2093.79) | 4834.0 (2946.12) | 10196.6 (6073.52) | 12665.3 (4808.41) | 19797.2 (10901.31)

5. Secondary Outcome: Poly Adenosine Diphosphate-ribose (PAR) Concentration in Peripheral Blood Monocyte or Mononuclear Cells of CEP-8983 (the Active Moiety of CEP-9722)
Time Frame: Predose (0 hour), 2 and 6 hours postdose on Days 1 and 15 of Cycle 1
Population: Pharmacodynamics was not evaluated in this study because the assay did not work due to sample collection methods.
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part 1: Overall Response Rate (ORR) - Percentage of Participants With the Best Tumor Response
Description: ORR was assessed by the best tumor response (complete response [CR], partial response [PR], stable disease [SD], and progressive disease [PD]) during the study using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). CR: Disappearance of all target and non-target lesions. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. PD: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions.
Time Frame: From the start of the treatment until disease progression/recurrence (up to 168 days)
Population: The safety analysis set included participants who received at least 1 dose of CEP-9722.
Measure: Number; unit: percentage of participants
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Number analyzed (Participants) | 3 | 7 | 8 | 6 | 5 | 6 | 9
percentage of participants | 67 | 71 | 75 | 83 | 80 | 50 | 56

7. Secondary Outcome: Part 2: Change in QT Interval
Time Frame: Day 1 and Day 15, Cycle 1
Population: Due to premature end of the study, Part 2 of the study was not conducted so there was no analysis of QT interval versus PK parameters.
Arm/Group | Overall Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first administration of CEP-9722 up 8 months
Description: The safety analysis set included participants who received at least 1 dose of CEP-9722.
Arm/Group | CEP-9722 Dose 1 QD | CEP-9722 Dose 1 BID | CEP-9722 Dose 2 BID | CEP-9722 Dose 3 BID | CEP-9722 Dose 4 BID | CEP-9722 Dose 5 BID | CEP-9722 Dose 6 BID
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/7 | 1/8 | 3/6 | 2/5 | 3/6 | 4/9
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 8/8 | 6/6 | 5/5 | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-9722 Dose 1 QD (N=3) | CEP-9722 Dose 1 BID (N=7) | CEP-9722 Dose 2 BID (N=8) | CEP-9722 Dose 3 BID (N=6) | CEP-9722 Dose 4 BID (N=5) | CEP-9722 Dose 5 BID (N=6) | CEP-9722 Dose 6 BID (N=9)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incoherent (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-9722 Dose 1 QD (N=3) | CEP-9722 Dose 1 BID (N=7) | CEP-9722 Dose 2 BID (N=8) | CEP-9722 Dose 3 BID (N=6) | CEP-9722 Dose 4 BID (N=5) | CEP-9722 Dose 5 BID (N=6) | CEP-9722 Dose 6 BID (N=9)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 4 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (5) | 3 (8) | 2 (3) | 3 (6) | 6 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (6) | 4 (9) | 3 (3) | 2 (2) | 8 (11)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 3 (7) | 2 (3) | 3 (3) | 8 (10)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device malfunction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (5) | 3 (3) | 5 (5) | 6 (7)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbohydrate antigen 125 increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (5) | 1 (1) | 4 (4) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedematous kidney (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to the reasons which are related to the pharmaceutical properties of the compound and not related to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.